CLINICAL TRIAL: NCT00612287
Title: Sublingual Buprenorphine for Chronic Pain in Patients at Risk for Drug Abuse
Brief Title: Sublingual Buprenorphine for Chronic Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Beth Israel Medical Center (Other)
Responsible Party: Andrew Rosenblum, PhD, National Development and Research Institutes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DA022675 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Pain
Keywords: Pain; Chronic pain; Buprenorphine; Drug addiction
MeSH Terms: conditions — Chronic Pain; Pain; Substance-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — Sublingual buprenorphine; product name Suboxone® (buprenorphine/naloxone). Dosing is informed by a clinical guideline which permits flexibility dependent up physician's clinical judgment. During the induction period (Day 1, at the physician's office) the first dose is 2 mg and can be brought up to 20 mg depending on patient's response. On Day 2 going forward dose can range from 2 mg q8h to 12 mg q8h. Rescue doses with buprenorphine are also permitted.
  Other Names: Suboxone®

SUMMARY:
The purpose of this study is to develop and pilot test clinical guidelines for the use of buprenorphine for the treatment chronic pain among patients with substance abuse histories. Buprenorphine, an opioid medication, holds promise as a treatment of chronic pain because, compared to most other opioid analgesics, it has a high safety profile, a low level of physical dependence, and mild withdrawal symptoms on cessation. Moreover there are promising reports from Europe of its use as a skin patch to treat chronic pain as well as clinical reports in the U.S. that it may be effective when used sublingually (placed under the tongue). This study will test the sublingual formulation.

ELIGIBILITY:
Inclusion Criteria:

Undergoing treatment for moderate-severe chronic pain for at least six months at either an ambulatory practice of the Department of Pain and Palliative Medicine Beth Israel Medical Center in New York City or the the Peter Kruger Clinic at the same institution.

Either

1. On opioid therapy (any dose) and observed to have had at least four of the aberrant drug-related behaviors described in (Passik et al. Clin J Pain; 22(2):173-81 2006) during the past six months, or
2. Considered a candidate for long-term therapy by the pain specialist and a history of a substance use disorder, as determined by DSM-IV criteria, but no longer meeting criteria for at least one year.

Age 18-70

Exclusion Criteria:

* Meets DSM-IV criteria for current opioid dependence or other substance use disorder including alcohol abuse.
* Currently being treated for opioid dependence with methadone.
* Currently maintained on naltrexone (e.g., for alcohol dependence).
* Taking benzodiazepines on a daily basis.
* A history of moderate-severe cardiopulmonary disease or symptoms or signs consistent with moderate-severe cardiopulmonary disease.
* Elevated liver function test (LFT) results (> 2.5 above normal).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-05 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 1, 2, 3, 4, 5 & 6 months

SECONDARY OUTCOMES:
Pain behaviors, psychiatric distress, drug use, side effects | Months 1 through 6

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenblum, PhD, Principal Investigator — NDRI
Locations (1):
- Beth Israel Medical Center, New York, New York, United States